CLINICAL TRIAL: NCT06603389
Title: The Development of Psychiatric Non-Suicidal Self-Injury Risk Assessment Scale (PNSSI-RAS)
Brief Title: The Development of Psychiatric Non-Suicidal Self-Injury Risk Assessment Scale
Status: Completed | Type: Observational
Sponsor: Shantou University Medical College (Other)
Responsible Party: Principal Investigator, Tang Hao, Master of Nursing Specialist, Shantou University Medical College
Other Study IDs: 202305
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Non Suicidal Self Injury
Keywords: Non-Suicidal Self-Injury; Risk Assessment; Scale development; Delphi method; Reliability; Validity; Nursing
MeSH Terms: conditions — Self-Injurious Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observation Group: Scales are used to get primary indicator and secondary indicators. The sample size should be set at 5 to 10 times the number of items, with a minimum total sample of 200. Additionally, an extra sample should be calculated to account for a potential 10-20% attrition rate, mitigating the impact of possible data loss. Given that the initial version scale consisted of 55 items, the minimum required sample size is 330.
  Interventions: Other: Psychiatric Non-Suicidal Self-Injury Risk Assessment Scale

INTERVENTIONS:
Other: Psychiatric Non-Suicidal Self-Injury Risk Assessment Scale — sacles or questionnaires

SUMMARY:
Non-suicidal self-injury (NSSI) is a growing global mental health challenge, distinct from suicidal behavior, with unique risk factors and mechanisms. Existing risk assessment tools do not focus on differentiating NSSI from suicidal self-harm or comprehensively evaluate risk and protective factors specific to NSSI. There is a lack of clinically applicable, validated scales dedicated to assessing NSSI risk, particularly in psychiatric populations. The present study is made to design the Psychiatric Non-Suicidal Self-Injury Risk Assessment Scale, a 39-item scale that evaluates static/dynamic risk factors and protective factors for NSSI in psychiatric patients.

DETAILED DESCRIPTION:
The initial item pool was created through literature review, semi-structured interviews, and group discussions. Two rounds of the Delphi were employed with twenty experts. We analyzed items using critical ratio, correlation coefficient, factor analysis, and Cronbach's α coefficient. Exploratory factor analysis determined item weights, while reliability analyses evaluated internal consistency, test-retest, inter-observer and split-half methods. In the validity analyses, CVI, construct validity and criterion validity were used. ROC curve established the optimal diagnostic threshold and the risk stratification was performed.

ELIGIBILITY:
Inclusion Criteria:

1. Criteria for inclusion in the sample were individuals , diagnosed with various mental disorders according to the International Classification of Diseases, 10th Revision (ICD-10) diagnostic criteria;
2. Gender is not limited and aged is 12-30 years old;
3. The patient's clinical profile is complete and the medical history is detailed;
4. Informed consent from patients or guardians who signed a consent for.

Exclusion Criteria:

The patient's clinical profile was incomplete and her medical history was not detailed.

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study, conducted between March and October 2023 at Shantou University Mental Health Center, enrolled 330 patients.
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2024-05-28 (Actual)

PRIMARY OUTCOMES:
Delphi Expert Consultation | Up to 8 weeks
  Two rounds of Delphi consultation were conducted with twenty experts who had a bachelor's degree or higher, senior titles, and more than ten years of experience in clinical psychiatry, nursing, or education. The experts rated the importance of each issue on a Likert scale (1: strongly disagree to 5: strongly agree) and made appropriate change suggestions.
  1. The authority coefficient (Cr) describes the expert's authority, and a value greater than 0.7 is deemed reliable. The formula is Cr=(Ca + Cs)/2;
  2. Kendall's coefficient of co-ordination (Kendall's W) and a chi-square test were used to assess expert opinion coordination, with statistical significance at p < 0.05;
  3. Item screening criteria include a mean item importance assignment of ≥ 3.50 and CV of ≤ 0.25. Expert opinions are combined to determine the scale's items;
  4. The questionnaire's recovery rate serves as a gauge for the experts' motivation.
Reliability | Through study completion, an average of 1 year
  The reliability was assessed using Cronbach α, test-retest reliability, inter-observer reliability, and split-half reliability methods. (1)Internal consistency: The higher the Cronbach α coefficient, the greater the reliability of the scale internal consistency.Cronbach α ≥ 0.9 indicates very good reliability, while 0.8 ≤ Cronbach α< 0.9 indicates high reliability. Cronbach α above 0.6 indicates adequate reliability; (2) Test-retest reliability: The closer the retest correlation coefficient tends to 1, the higher the retest reliability; (3)Inter-observer reliability: Inter-rater reliability approaches 1, signifying greater reliability of the scale. Inter-rater reliability should be at least > 0.6, and > 0.75 indicates that the scale possesses relatively high reliability. (4)Split-half reliability: Split-half reliability coefficients greater than 0.70 for the scale as a whole and for each dimension are widely regarded as good.
Validity | Through study completion, an average of 1 year
  1. CVI: The I-CVI was the number of experts who rated 4-5 divided by the total number of experts; the S-CVI was separated into two parts: S-CVI/Ave and S-CVI/Ua; I-CVI > 0.78 and S-CVI ≥ 0.9 indicate strong content validity；
  2. Construct validity: The maximum variance approach was used in exploratory factor analysis to extract KMO values, Bartlett's test of sphericity values, component matrix (factor loading values), initial eigenvalues, percentage of variance for each component, and cumulative variance contribution ratio;
  3. Criterion validity: The Barrett Impulsivity Scale (BIS-11) was used as a validity scale to assess the validity of the scale's correlational validity. The higher the correlation coefficient, the better the validity.
Diagnostic Thresholds | Up to 2 weeks.
  The Receiver Operator Characteristic (ROC) was used to characterize the subject and the maximum value of the Youden Index (YI) was used as a threshold to find the optimal diagnostic threshold.
Risk Stratification | Up to 2 weeks.
  Based on the optimal diagnostic threshold, true-positive patients were screened and the degree of risk of non-suicidal self-harm in patients with mental disorders was graded using the interquartile method, defining P0-P25 as grade I, P25-P75 as grade II, and P75-P100 as grade III.

SECONDARY OUTCOMES:
The Barratt Impulsiveness Scale (BIS-11) | Through study completion, an average of 1 year
  Criterion validity. The 30 items in the revised Chinese version of the Barratt Impulsivity Scale are divided into three categories: Motor Impulsivity, Cognitive Impulsiveness and Non-Planning Impulsiveness. Each item is scored on a Likert scale (not, rarely, sometimes, often, always), with the Planning and Cognitive subscales reverse scored and the Motor subscale positive. The total scores range from 30 to 150, with higher scores denoting higher levels of impulsivity and high scores on the three subscales representing hyperactivity, inattention, and lack of planning.

CONTACTS AND LOCATIONS:
Overall Officials: Jingfang Chen, Bachelor, Study Director — Shantou University Mental Health Center
Locations (1):
- Shantou University Mental Health Center, Shantou, Guangdong, China